CLINICAL TRIAL: NCT01671982
Title: Tenofovir Pharmacokinetics in HIV-infected Thai Adults With Moderate Renal Function Impairment Receiving Either a Non-nucleoside Reverse Transcriptase Inhibitor (NNRTI)-Based or Lopinavir/Ritonavir-based Antiretroviral Therapy
Brief Title: ALternative TEnofovir Dosing in Adults With Moderate Renal Function Impairment
Acronym: ALTER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: The Government Pharmaceutical Organization (Other Government); Chiang Mai University (Other)
Responsible Party: Principal Investigator, GONZAGUE JOURDAIN, Researcher, Institut de Recherche pour le Developpement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER
Record Dates: First submitted 2012-08-17; First posted 2012-08-24 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tenofovir-containing HAART (Experimental)
  Interventions: Other: Tenofovir Dose Adjustment

INTERVENTIONS:
Other: Tenofovir Dose Adjustment — In subjects with a confirmed CLcr 30 to <50 mL/min, switch tenofovir 300 mg every 48 hours, to 150 mg once daily for 2 weeks.

SUMMARY:
To assess the drug concentrations of tenofovir (TDF) in HIV-infected Thai adults with moderate renal function impairment when administered at the recommended dose of 300 mg every 48 hours, and at an alternative dose of 150 mg every 24 hours.

DETAILED DESCRIPTION:
The study is designed as a Phase I, non-randomized, open-label, pharmacokinetic study. We hypothesize that administration of tenofovir 150 mg once daily to HIV-infected Thai adults with moderate renal function impairment (CLcr between 30 to <50 mL/min) will provide comparable drug exposure to the current recommended dose of 300 mg every 48 hours.

Confirmed HIV-positive subjects receiving tenofovir (TDF) 300 mg, every 48 hours, as part of an NNRTI-based or lopinavir/ritonavir (LPV/r)-based HAART regimen will be proposed to participate.

Subjects meeting the required criteria will be enrolled into one of 2 groups depending on their HAART regimen: .

Group 1: Subjects receiving tenofovir 300 mg, every 48 hours, in combination with lamivudine and an NNRTI,and a confirmed CLcr 30 to <50 mL/min

Group 2: Subjects receiving tenofovir 300 mg, every 48 hours, in combination with lamivudine and lopinavir/ritonavir, and a confirmed CLcr 30 to <50 mL/min

The study procedures are identical for both groups. All subjects enrolled will have two study visits. At the first visit, a 48-hour pharmacokinetic evaluation will be performed. Immediately following completion of the PK sampling, the tenofovir dose will be changed to 150 mg, once daily. Two weeks later, at the second visit, a 24-hour pharmacokinetic evaluation will be performed. Following completion of the second PK sampling the tenofovir dose will be changed back to 300 mg every 48 hours. At this time the subjects has reach the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old
* provided written informed consent
* receiving the tenofovir tablet formulation from the Thai Government Pharmaceutical Organization (GPO) for at least 4 weeks before enrollment
* documentation of confirmed HIV-1 infection (documented by two serology tests obtained at two different dates)
* Confirmed Creatinine clearance result between 30 to <50 mL/min [confirmed defined as two CLcr determinations calculated using the Cockcroft-Gault equation within two weeks of each other, within 1 month prior to entry]
* received tenofovir 300 mg, every 48 hours for at least 2 weeks prior to entry, in combination with 3TC plus NNRTI, or 3TC plus lopinavir/ritonavir
* a HIV-1 RNA viral load < 50 copies/mL within 6 months prior to entry

Exclusion Criteria:

* Concomitant use of a atazanavir, didanosine
* Pregnant
* Any of the following laboratory tests within 30 days prior to study entry classified as ≥ Grade 3 (see DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0 [Dec. 2004], Clarification August, 2009): neutrophil count, hemoglobin, platelets, AST, or ALT
* HBs-antigen positive
* Any clinically significant diseases (other than HIV-1 infection) or clinically significant findings during the screening medical history or physical examination that, in the investigator's opinion, would compromise participation in this study
* concurrent participation to any other clinical trial without prior agreement of the two study teams

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2014-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Tenofovir plasma area-under the concentration time curve (AUC) | Study Entry and Day 14
  For each patient, ratios of AUC0-last of q24h versus q48h will be calculated. Geometric mean ratios (GMRs) with 90% CI will be calculated after log-transformation of within patient ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Tim R Cressey, PhD, Principal Investigator — PHPT / Chiang Mai University / IRD
Locations (5):
- Thailand (5):
  - Chonburi Hospital, Chon Buri, Changwat Chon Buri
  - Sanpatong Hospital, Sanpatong, Chiang Mai
  - HIV-NAT, Bangkok
  - Nakornping Hospital, Chiang Mai
  - Phayao Hospital, Phayao

REFERENCES:
- [Result] Cressey TR, Avihingsanon A, Halue G, Leenasirimakul P, Sukrakanchana PO, Tawon Y, Jaisieng N, Jourdain G, Podany AT, Fletcher CV, Klinbuayaem V, Bowonwatanuwong C. Plasma and Intracellular Pharmacokinetics of Tenofovir Disoproxil Fumarate 300 mg Every 48 Hours vs 150 mg Once Daily in HIV-Infected Adults With Moderate Renal Function Impairment. Clin Infect Dis. 2015 Aug 15;61(4):633-9. doi: 10.1093/cid/civ346. Epub 2015 Apr 28. PMID 25921689
- See also: Related Info — http://www.phpt.org